CLINICAL TRIAL: NCT00808652
Title: Prevalence and Outcome of Brachial Artery Endothelial Function in Morbidly Obese Patients Undergoing Bariatric Surgery
Status: Terminated | Type: Observational
Why Stopped: not enough recruits
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-5431-08-DG-CTIL
Record Dates: First submitted 2008-12-12; First posted 2008-12-16 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Obesity, Morbid; Ischemic Heart Disease
MeSH Terms: conditions — Obesity, Morbid; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Measurement of flow mediated dilation of brachial artery. — Flow-mediated brachial artery reactivity will be measured and flow-mediated vasodilatation will be assessed with the subject's arm using a 15 MHz linear array ultrasound.
  Study Phases:
  1. Flow-mediated (endothelial-dependent) vasodilatation (FMD): Following a 2-minute baseline period, a longitudinal image of the artery will be obtained. A tourniquet placed around the forearm proximal to the target artery will be inflated to a pressure 50 mmHg higher than the subject's systolic blood pressure and held for 5 minutes. Cuff will be then deflated. A continuous scan will be performed at deflation, 60 and 90 seconds after cuff deflation, with frozen and Doppler measurements recorded at similar intervals to the baseline phase.
  2. NTG-induced (non-endothelial-dependent) vasodilatation (NTG): After vessel recovery, sublingual 375 mg of isosorbide dinitrate spray will be administered, and scanning will be performed continuously for 5 minutes thereafter.

SUMMARY:
The relation between obesity and ischemic heart disease (IHD) is under considerable debate. The reduction in all-cause mortality and, more specifically, the reduction in cardiac-related mortality seen after weight-loss surgery, may be due to regression or slowing developement of subclinical IHD. Function of cells lining the arteries (endothelium) is closely related to the state of IHD and its measurement can serve as a surrogate marker for the existence and severity of IHD. The investigators hypothesize that the prevalence of undiagnosed IHD in the morbidly obese population is high and that following surgery for weight reduction there is a halt in the progression, or even a regression in its severity.

The study includes measurement of endothelial function before and after weight-reducing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients who fulfill the NIH criteria for surgical intervention.

Exclusion Criteria:

* Patients deemed unfit for surgery
* Pregnant women, or who are attempting conception.
* Subjects with any history of myocardial infarction, coronary artery bypass grafting surgery, coronary angiography with angioplasty and/or stenting, or any lesion > 50% of the coronary artery luminal diameter, cerebrovascular accident, or peripheral vascular disease with abnormal electrocardiograms and/or echocardiography.
* History of drug or alcohol abuse.
* Chronic liver disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbisly obese patients scheduled to undergo bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2009-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Flow-mediated (endothelial-dependent) vasodilatation (FMD) difference (before vs after surgery) | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No